CLINICAL TRIAL: NCT03039192
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Adult Subjects Assessed to be at Imminent Risk for Suicide
Brief Title: 54135419SUI3001: A Study to Evaluate the Efficacy and Safety of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Adult Participants Assessed to be at Imminent Risk for Suicide
Acronym: Aspire I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108284; 2016-003990-17 (EudraCT Number); 54135419SUI3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Esketamine + Standard of care (Experimental): Participants will receive intranasal esketamine 84 milligram (mg) two times per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25) along with standard of care (SOC) antidepressant treatment.
  Interventions: Drug: Esketamine; Other: Standard of Care
- Placebo + Standard of care (Placebo Comparator): Participants will receive intranasal placebo two times per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25) along with standard of care antidepressant treatment.
  Interventions: Other: Placebo; Other: Standard of Care

INTERVENTIONS:
Drug: Esketamine — Intranasal esketamine solution 84 milligram (mg)
  Arms: Esketamine + Standard of care
Other: Placebo — Intranasal Placebo solution
  Arms: Placebo + Standard of care
Other: Standard of Care — The standard of care antidepressant treatment (antidepressant monotherapy or antidepressant plus augmentation therapy) will be determined by the treating physician(s) based on clinical judgement and practice guidelines prior to randomization, and the treatment will be initiated on Day 1.

SUMMARY:
The purpose of the study is to evaluate the efficacy of intranasal esketamine 84 milligram (mg) compared with intranasal placebo in addition to comprehensive standard of care in reducing the symptoms of Major Depressive Disorder (MDD), including suicidal ideation, in participants who are assessed to be at imminent risk for suicide, as measured by the change from baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) total score at 24 hours post first dose.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance which contains no drug) that is compared in a clinical trial with a drug to test if the drug has a real effect), multicenter (when more than one hospital or study team work on a medical research study) study. Study will enroll participants with suicidal ideation who are assessed to be at imminent risk for suicide. The study will consist of a screening evaluation performed within 48 hours prior to the Day 1 intranasal dose immediately followed by a 25-day double-blind treatment phase (Day 1 to 25), and a 65 day follow-up phase (Day 26 to Day 90). The total study duration for each subject will be approximately 13 weeks. Participants' safety will be evaluated throughout the study. If you or a loved one are having thoughts of suicide, please seek immediate medical help. Go to the emergency room or call the National Suicide Prevention Lifeline at 1-800-273-8255.

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) diagnostic criteria for Major Depressive Disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Mini International Psychiatric Interview (MINI)
* In the physician's opinion, acute psychiatric hospitalization is clinically warranted due to participant's imminent risk of suicide
* Participants must have current suicidal ideation with intent, confirmed by a "Yes" response to Question B3 [Think (even momentarily) about harming or of hurting or of injuring yourself: with at least some intent or awareness that you might die as a result; or think about suicide (ie, about killing yourself)?] and Question B10 [Intend to act on thoughts of killing yourself?] obtained from the MINI. Note: the response to B3 must refer to the present, whereas the response to B10 may reflect the past 24 hours. If the screening period is longer than 24 hours, assessment of B3 and B10 of MINI must be repeated prior to randomization to confirm eligibility
* Participant has a Montgomery Asberg Depression Rating Scale (MADRS) total score of greater than (>) 28 predose on Day 1
* As part of standard of care treatment, participant agrees to be hospitalized voluntarily for a recommended period of 5 days after randomization (may be shorter or longer if clinically warranted in the investigator's opinion) and take prescribed non-investigational antidepressant therapy(ies) for at least the duration of the double-blind treatment phase (Day 25)
* Participant is comfortable with self-administration of intranasal medication and able to follow instructions provided

Exclusion Criteria:

* Participant has a current DSM-5 diagnosis of bipolar (or related disorders), antisocial personality disorder, or obsessive compulsive disorder
* Participant currently meets DSM-5 criteria for borderline personality disorder. Participant not meeting full DSM-5 criteria for borderline personality disorder but exhibiting recurrent suicidal gestures, threats, or self-mutilating behaviors should also be excluded
* Participant has a current clinical diagnosis of autism, dementia, or intellectual disability
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder, or MDD with psychotic features
* Participant meets the DSM-5 severity criteria for moderate or severe substance or alcohol use disorder, (except for nicotine or caffeine), within the 6 months before screening. A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (56):
- United States (17):
  - UAB Department of Psychiatry and Behavioral Neurobiology, Birmingham, Alabama
  - Metropolitan Neuro Behavioral Institute, Chandler, Arizona
  - Collaborative NeuroScience Network, Garden Grove, California
  - Yale University, New Haven, Connecticut
  - Rush University, Chicago, Illinois
  - Alexian Behavioral Health Hospital, Hoffman Estates, Illinois
  - University of Louisville Department of Psychiatry, Louisville, Kentucky
  - LSU Health Sciences Center New Orleans, New Orleans, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - State University of New York, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Clinical Trials of America, Hickory, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Bulgaria (5):
  - Regional Psychiatric Dispansery, Bulgaria
  - Mental Health Center Prof. Dr. Ivan Temkov, Burgas
  - State Psychiatric Hospital - Lovech, Lovech
  - UMHAT 'Sveti Georgi'-Plovdiv, Plovdiv
  - Military Medical Academy Multiprofile Hospital for Active Treatment Sofia, Sofia
- Estonia (2):
  - North Estonian Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Germany (3):
  - Vivantes Humboldt Klinikum, Berlin
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Klinik für Psychiatrie und Psychotherapie, Freiburg im Breisgau
- Hungary (5):
  - Eszak Kozep budai Centrum Uj Szent Janos Korhaz es Szakrendelo Budai Csaladkozpontu, Budapest
  - Semmelweis Egyetem Kútvölgyi Klinikai Tömb, Budapest
  - Nyiro Gyula Korhaz, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Malaysia (4):
  - University Kebangsaan Malaysia Medical Centre, Cheras
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tuanku Jaafar, Seremban
- Fakultna nemocnica s poliklinikou v Ziline, Žilina, Slovakia
- South Africa (2):
  - Flexivest 14 Research, Cape Town
  - Juan Schrönen - Western Cape South Africa, Welgemoed
- South Korea (5):
  - Chonnam National University Hospital, Gwangju
  - Korea University Ansan Hospital, Gyeonggi-do
  - Kyung Hee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (8):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Internac. Neurociencias Aplicadas, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Benito Menni Comp. Asist. Salut Mental, Sant Boi de Llobregat
- Taiwan (4):
  - Tri-Service Genaral Hospital, Neihu District
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Fu DJ, Zhang Q, Shi L, Borentain S, Guo S, Mathews M, Anjo J, Nash AI, O'Hara M, Canuso CM. Esketamine versus placebo on time to remission in major depressive disorder with acute suicidality. BMC Psychiatry. 2023 Aug 11;23(1):587. doi: 10.1186/s12888-023-05017-y. PMID 37568081
- [Derived] Jamieson C, Canuso CM, Ionescu DF, Lane R, Qiu X, Rozjabek H, Molero P, Fu DJ. Effects of esketamine on patient-reported outcomes in major depressive disorder with active suicidal ideation and intent: a pooled analysis of two randomized phase 3 trials (ASPIRE I and ASPIRE II). Qual Life Res. 2023 Nov;32(11):3053-3061. doi: 10.1007/s11136-023-03451-9. Epub 2023 Jul 13. PMID 37439961
- [Derived] Turkoz I, Lopena O, Salvadore G, Sanacora G, Shelton R, Fu DJ. Treatment response to esketamine nasal spray in patients with major depressive disorder and acute suicidal ideation or behavior without evidence of early response: a pooled post hoc analysis of ASPIRE. CNS Spectr. 2023 Aug;28(4):482-488. doi: 10.1017/S1092852922000931. Epub 2022 Jul 29. PMID 35904046
- [Derived] Rozjabek H, Li N, Hartmann H, Fu DJ, Canuso C, Jamieson C. Assessing the meaningful change threshold of Quality of Life in Depression Scale using data from two phase 3 studies of esketamine nasal spray. J Patient Rep Outcomes. 2022 Jul 10;6(1):74. doi: 10.1186/s41687-022-00453-y. PMID 35816217
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Canuso CM, Ionescu DF, Li X, Qiu X, Lane R, Turkoz I, Nash AI, Lopena TJ, Fu DJ. Esketamine Nasal Spray for the Rapid Reduction of Depressive Symptoms in Major Depressive Disorder With Acute Suicidal Ideation or Behavior. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):516-524. doi: 10.1097/JCP.0000000000001465. PMID 34412104
- [Derived] Fu DJ, Ionescu DF, Li X, Lane R, Lim P, Sanacora G, Hough D, Manji H, Drevets WC, Canuso CM. Esketamine Nasal Spray for Rapid Reduction of Major Depressive Disorder Symptoms in Patients Who Have Active Suicidal Ideation With Intent: Double-Blind, Randomized Study (ASPIRE I). J Clin Psychiatry. 2020 May 12;81(3):19m13191. doi: 10.4088/JCP.19m13191. PMID 32412700
- See also: A Study to Evaluate the Efficacy and Safety of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation (Aspire I) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108284&attachmentIdentifier=0b008702-9e7b-4d11-b853-d3aba96bb3a1&fileName=54135419SUI3001_(CR108284)_Additional_Results_Data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Plus SOC Antidepressant Treatment: Participants self-administered placebo matched to esketamine intranasally (1 spray of placebo to each nostril at 0, 5 and 10 minutes) twice per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25) plus received standard of care (SOC) antidepressant treatment which was initiated or optimized on Day 1.
- Esketamine 84 mg Plus SOC Antidepressant Treatment: Participants self-administered esketamine 84 milligrams (mg) intranasally (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) twice per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25) and received SOC antidepressant treatment which was initiated or optimized on Day 1.
Period: Overall Study
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Started | 112 | 114
Treated | 112 | 113
Completed | 80 | 84
Not Completed | 32 | 30
Not completed — Lost to Follow-up | 4 | 4
Not completed — Adverse event, serious fatal | 0 | 1
Not completed — Adverse event, non-fatal | 0 | 2
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Discontinued from treatment phase | 19 | 12
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study agent in the double-blind treatment phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment | Total
Number analyzed (Participants) | 112 | 113 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (12.54) | 40.8 (13.11) | 39.3 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 66 | 139
  Male | 39 | 47 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 28 | 28 | 56
  Black or African American | 7 | 5 | 12
  More than one race | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 2 | 1 | 3
  White | 74 | 77 | 151
Region of Enrollment [Count of Participants; unit: Participants]
  BULGARIA | 10 | 9 | 19
  ESTONIA | 1 | 3 | 4
  GERMANY | 10 | 8 | 18
  HUNGARY | 8 | 7 | 15
  MALAYSIA | 9 | 7 | 16
  SOUTH AFRICA | 8 | 7 | 15
  SOUTH KOREA | 10 | 10 | 20
  SPAIN | 20 | 24 | 44
  TAIWAN | 8 | 9 | 17
  UNITED STATES | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at 24 Hours After the First Dose (Day 2) (Last Observation Carried Forward [LOCF] Data) During Double-blind Phase
Description: MADRS is clinician-rated scale designed to be used in participants with Major Depressive Disorder (MDD) to measure depression severity and detect changes due to antidepressant treatment. It evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic and suicidal thoughts. Scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms), summed for total possible score of 0 to 60. Higher scores represent more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1, predose) and 24 hours first post dose (Day 2)
Population: Full efficacy analysis set included all randomized participants who received at least 1 dose of intranasal study agent during double-blind phase and have had both a baseline and a postbaseline evaluation for MADRS total score or CGI-SS-R. Here, N (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 111
units on a scale | -12.8 (10.73) | -16.4 (11.95)
Statistical Analysis 1: Comparison: Placebo Plus SOC Antidepressant Treatment vs Esketamine 84 mg Plus SOC Antidepressant Treatment; Test type: Superiority; p = 0.006, ANCOVA; Difference of Least Square Means = -3.8, 95% CI 2-sided [-6.56 to -1.09], Standard Error of Mean 1.39

2. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity of Suicidality- Revised (CGI-SS-R) Score at 24 Hours After the First Dose (Day 2) (LOCF Data) During Double-blind Phase
Description: CGI-SS-R was derived from the Clinical Global Impression Severity Scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participants illness. The CGI-SS-R rating is scored on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants). A higher score indicates a more severe condition and a reduction in score indicates improvement (that is, lower severity of suicidality).
Time Frame: Baseline (Day 1, predose) and 24 hours first post dose (Day 2)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 111
units on a scale | -1.0 [-5 to 1] | -1.0 [-6 to 2]

3. Secondary Outcome: Number of Participants Who Achieved Remission (MADRS Total Score Less Than or Equal to [<=] 12) Through the Double-blind Phase
Description: Participants who had a MADRS total score of <=12 were considered remitters. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition and a negative change in score indicates improvement.
Time Frame: Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and Day 25 (predose and 4 hours postdose)
Population: Full efficacy analysis set included all randomized participants who received at least 1 dose of intranasal study agent during the double-blind phase and have had both a baseline and a post-baseline evaluation for the MADRS total score or CGI-SS-R.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
Participants
  Day 1 (4 Hours postdose) | 9 | 12
  Day 2 | 10 | 21
  Day 4 | 13 | 28
  Day 8 | 23 | 30
  Day 11 | 26 | 33
  Day 15 | 29 | 38
  Day 18 | 30 | 42
  Day 22 | 25 | 41
  Day 25 (Predose) | 38 | 46
  Day 25 (4 hours postdose) | 42 | 60

4. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale Total Score at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25 During Double-blind Phase
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition and a negative change in score indicates improvement.
Time Frame: Baseline and Days 1, 2, 4, 8, 11, 15, 18, 22 and 25 (predose and 4 hours postdose)
Population: Full efficacy analysis set included all randomized participants who received at least 1 dose of intranasal study agent during double-blind phase and have had both a baseline and a post-baseline evaluation for MADRS total score or CGI-SS-R. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 1: number analyzed (Participants) | 112 | 110
  Change at Day 1 | -10.9 (9.69) | -13.5 (10.89)
  Change at Day 2: number analyzed (Participants) | 111 | 111
  Change at Day 2 | -12.9 (10.72) | -16.4 (11.95)
  Change at Day 4: number analyzed (Participants) | 110 | 109
  Change at Day 4 | -14.5 (11.39) | -19.1 (12.29)
  Change at Day 8: number analyzed (Participants) | 108 | 104
  Change at Day 8 | -17.4 (12.59) | -19.7 (12.91)
  Change at Day 11: number analyzed (Participants) | 103 | 100
  Change at Day 11 | -19.0 (12.08) | -21.8 (12.20)
  Change at Day 15: number analyzed (Participants) | 99 | 104
  Change at Day 15 | -20.4 (12.19) | -22.3 (11.70)
  Change at Day 18: number analyzed (Participants) | 94 | 102
  Change at Day 18 | -21.4 (12.00) | -23.9 (11.77)
  Change at Day 22: number analyzed (Participants) | 92 | 103
  Change at Day 22 | -21.6 (12.32) | -24.0 (12.38)
  Change at Day 25: predose: number analyzed (Participants) | 92 | 96
  Change at Day 25: predose | -23.0 (12.41) | -24.8 (13.63)
  Change at Day 25 (4 hours postdose): number analyzed (Participants) | 88 | 94
  Change at Day 25 (4 hours postdose) | -25.8 (10.94) | -29.5 (10.89)

5. Secondary Outcome: Change From Baseline in Clinical Global Impression- Severity of Suicidality-Revised (CGI-SS-R) at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25 During Double-blind Phase
Description: CGI-SS-R was derived from the Clinical Global Impression Severity Scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participants illness. The CGI-SS-R rating is scored on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants). A higher score indicates a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline and Days 1, 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 1: number analyzed (Participants) | 112 | 110
  Change at Day 1 | 0.0 [-5 to 1] | -1.0 [-6 to 1]
  Change at Day 2 | -1.0 [-5 to 1] | -1.0 [-6 to 2]
  Change at Day 4: number analyzed (Participants) | 110 | 110
  Change at Day 4 | -1.0 [-5 to 1] | -2.0 [-6 to 2]
  Change at Day 8: number analyzed (Participants) | 108 | 105
  Change at Day 8 | -2.0 [-5 to 0] | -2.0 [-6 to 1]
  Change at Day 11: number analyzed (Participants) | 102 | 101
  Change at Day 11 | -2.0 [-5 to 1] | -3.0 [-6 to 1]
  Change at Day 15: number analyzed (Participants) | 99 | 105
  Change at Day 15 | -2.0 [-5 to 0] | -3.0 [-5 to 0]
  Change at Day 18: number analyzed (Participants) | 94 | 103
  Change at Day 18 | -2.5 [-5 to 0] | -3.0 [-6 to 1]
  Change at Day 22: number analyzed (Participants) | 91 | 105
  Change at Day 22 | -3.0 [-5 to 1] | -3.0 [-6 to 1]
  Change at Day 25: number analyzed (Participants) | 93 | 96
  Change at Day 25 | -3.0 [-5 to 1] | -3.0 [-6 to 1]

6. Secondary Outcome: Number of Participants Who Achieved Resolution of Suicidality (CGI-SS-R Score of 0 or 1) Through Double-blind Phase
Description: CGI-SS-R was derived from the Clinical Global Impression Severity Scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participants illness. The CGI-SS-R rating is scored on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants). A higher score indicates a more severe condition. Negative change in score indicates improvement. A participant was considered to achieve resolution of suicidality at a given time point if the CGI-SS-R score was 0 (normal, not at all suicidal) or 1 (questionably suicidal).
Time Frame: Days 1, 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
Participants
  Day 1 | 25 | 37
  Day 2 | 39 | 42
  Day 4 | 45 | 49
  Day 8 | 48 | 53
  Day 11 | 46 | 60
  Day 15 | 52 | 68
  Day 18 | 55 | 68
  Day 22 | 62 | 70
  Day 25 | 57 | 71

7. Secondary Outcome: Change From Baseline in Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) Scale Total Score at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25 During Double-blind Phase
Description: The CGI-SR-I is a scale summarizing the clinician's best assessment of the likelihood that the participant will attempt suicide in the next 7 days. The CGI-SR-I rating is scored on a 7-point scale: where' 0 (no imminent suicide risk); 1 (minimal imminent suicide risk), 2 (mild imminent suicide risk), 3 (moderate imminent suicide risk), 4 (marked imminent suicide risk), 5 (severely imminent suicide risk), 6 (extreme imminent suicide risk). Higher score indicates a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline and Days 1, 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 1: number analyzed (Participants) | 112 | 110
  Change at Day 1 | 0.0 [-4 to 2] | -1.0 [-5 to 3]
  Change at Day 2 | -1.0 [-5 to 2] | -1.0 [-5 to 2]
  Change at Day 4: number analyzed (Participants) | 110 | 110
  Change at Day 4 | -1.0 [-5 to 2] | -2.0 [-5 to 2]
  Change at Day 8: number analyzed (Participants) | 108 | 105
  Change at Day 8 | -2.0 [-5 to 2] | -2.0 [-6 to 1]
  Change at Day 11: number analyzed (Participants) | 102 | 101
  Change at Day 11 | -2.0 [-5 to 1] | -2.0 [-6 to 1]
  Change at Day 15: number analyzed (Participants) | 99 | 105
  Change at Day 15 | -2.0 [-5 to 2] | -3.0 [-5 to 2]
  Change at Day 18: number analyzed (Participants) | 94 | 103
  Change at Day 18 | -3.0 [-5 to 1] | -3.0 [-5 to 2]
  Change at Day 22: number analyzed (Participants) | 91 | 105
  Change at Day 22 | -3.0 [-5 to 1] | -3.0 [-6 to 1]
  Change at Day 25: number analyzed (Participants) | 93 | 96
  Change at Day 25 | -3.0 [-5 to 2] | -3.0 [-6 to 1]

8. Secondary Outcome: Change From Baseline in Beck Hopelessness Scale (BHS) Total Score at Days 8 and 25 During Double-blind Phase
Description: BHS is a self-reported measure to assess one's level of negative expectations or pessimism regarding future. It consists of 20 true-false items that examine respondent's attitude over past week by either endorsing a pessimistic statement or denying an optimistic statement; 9 are keyed false and 11 are keyed true. For every statement, each response was assigned score of 0 or 1. Total BHS score is sum of item responses, ranged from 0-20, where higher score represented higher level of hopelessness.
Time Frame: Baseline, Days 8 and 25
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 8: number analyzed (Participants) | 108 | 111
  Change at Day 8 | -4.4 (6.03) | -5.3 (6.06)
  Change at Day 25: number analyzed (Participants) | 98 | 105
  Change at Day 25 | -6.6 (6.63) | -6.9 (6.92)

9. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) at Days 2, 11 and 25 During Double-blind Phase: Health Status Index
Description: EQ-5D-5L measures health outcome. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). EQ-5D-5L system comprises following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of 5 dimensions is divided into 5 levels of perceived problems (Level 1-no problem, Level 2-slight problems, Level 3-moderate problems, Level 4-severe problems, Level 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a health status index (HSI). Health Status Index ranges from 0.148 - 0.949, anchored at 0 (dead) and 1 (full health). Positive change in score indicates improvement.
Time Frame: Baseline and Days 2, 11 and 25
Population: Full efficacy analysis set included all randomized participants who received at least 1 dose of intranasal study agent during double-blind phase, have had both a baseline and a post-baseline evaluation for MADRS total score or CGI-SS-R. Here, 'n' (number analyzed) signifies number of participants who were analyzed at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 2: number analyzed (Participants) | 110 | 111
  Change at Day 2 | 0.096 (0.1785) | 0.156 (0.1944)
  Change at Day 11: number analyzed (Participants) | 107 | 106
  Change at Day 11 | 0.169 (0.2139) | 0.206 (0.2043)
  Change at Day 25: number analyzed (Participants) | 97 | 104
  Change at Day 25 | 0.189 (0.2336) | 0.227 (0.2078)

10. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) at Days 2, 11 and 25 During Double-blind Phase: EQ-Visual Analogue Scale (EQ-VAS)
Description: EQ-5D-5L measures health outcome. It consists of EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ-VAS). EQ-VAS score from 0 (worst health) to 100 (best health), positive change in score indicates improvement.
Time Frame: Baseline, Days 2, 11 and 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 2: number analyzed (Participants) | 110 | 111
  Change at Day 2 | 7.8 (17.32) | 13.5 (20.78)
  Change at Day 11: number analyzed (Participants) | 107 | 106
  Change at Day 11 | 16.3 (22.27) | 17.9 (24.55)
  Change at Day 25: number analyzed (Participants) | 97 | 104
  Change at Day 25 | 20.0 (23.49) | 21.4 (26.71)

11. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) at Days 2, 11 and 25 During Double-blind Phase: Sum Score
Description: EQ-5D-5L measures health outcome. It consists of EQ-5D-5L system and EQ-VAS. EQ-5D-5L system comprises following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of 5 dimensions is divided into 5 levels of perceived problems (Level 1-no problem, Level 2-slight problems, Level 3-moderate problems, Level 4-severe problems, and Level 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a health status index (HSI). Health Status Index ranges from 0.148 - 0.949, anchored at 0 (dead) and 1 (full health), a lower score indicates worse health. Sum score=(sum of the scores from the 5 dimensions minus 5)*5. Sum score ranges from 0-100. Higher score indicates a more severe problem. Negative change in score indicates improvement.
Time Frame: Baseline, Days 2, 11 and 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 2: number analyzed (Participants) | 110 | 111
  Change at Day 2 | -6.1 (12.28) | -11.2 (14.87)
  Change at Day 11: number analyzed (Participants) | 107 | 106
  Change at Day 11 | -12.3 (16.23) | -15.2 (15.75)
  Change at Day 25: number analyzed (Participants) | 97 | 104
  Change at Day 25 | -13.4 (18.05) | -16.8 (16.30)

12. Secondary Outcome: Change From Baseline in Quality of Life in Depression Scale (QLDS) Total Score at Days 2, 11 and 25 During Double-blind Phase
Description: The QLDS is a disease specific patient-reported outcome designed to assess health related quality of life in participants with major depressive disorder (MDD). The instrument has a recall period of "at the moment", contains 34-items with "true"/"not true" response options and takes approximately 5-10 minutes to complete. The total score range is from 0 (good quality of life) to 34 (very poor quality of life). A higher score indicates a more severe condition. Negative change indicates improvement.
Time Frame: Baseline and Days 2, 11 and 25
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 2: number analyzed (Participants) | 110 | 112
  Change at Day 2 | -2.5 (4.55) | -3.1 (5.14)
  Change at Day 11: number analyzed (Participants) | 107 | 106
  Change at Day 11 | -4.4 (5.93) | -5.6 (5.92)
  Change at Day 25: number analyzed (Participants) | 97 | 104
  Change at Day 25 | -5.6 (5.99) | -6.8 (5.97)

13. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM-9) Total Score at Days 15 and 25 During Double-blind Phase
Description: The TSQM-9 is a 9-item generic patient-reported outcome instrument to assess participants' satisfaction with medication. It covers domains of effectiveness, convenience, and global satisfaction. The TSQM-9 domain scores were calculated as recommended by the instrument authors. (i) Effectiveness = [(item 1 + item 2 + item 3) - 3]/18*100, (ii) Convenience = [(item 4 + item 5 + item 6) - 3]/18*100 and (iii) Global satisfaction = [(item 7 + item 8 + item 9) - 3]/14*100. Each domain score can be calculated only if all the three items considered in the calculation of that score are not missing. The TSQM-9 domain score ranges from 0 to 100, with higher scores representing higher satisfaction.
Time Frame: Days 15 and 25
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Effectiveness: Day 15: number analyzed (Participants) | 105 | 108
  Effectiveness: Day 15 | 51.7 (25.74) | 63.5 (23.72)
  Effectiveness: Day 25: number analyzed (Participants) | 96 | 102
  Effectiveness: Day 25 | 57.6 (24.66) | 65.8 (25.23)
  Convenience: Day 15: number analyzed (Participants) | 105 | 108
  Convenience: Day 15 | 70.9 (19.57) | 70.5 (20.75)
  Convenience: Day 25: number analyzed (Participants) | 96 | 102
  Convenience: Day 25 | 74.0 (19.38) | 71.3 (19.69)
  Global Satisfaction: Day 15: number analyzed (Participants) | 105 | 108
  Global Satisfaction: Day 15 | 52.2 (28.57) | 64.5 (24.62)
  Global Satisfaction: Day 25: number analyzed (Participants) | 96 | 102
  Global Satisfaction: Day 25 | 55.7 (27.44) | 68.5 (25.51)

14. Secondary Outcome: Change From Baseline in Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 5 (My Risk) Question 3 (Patient-reported FoST) Total Score at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25 During Double-blind Phase
Description: SIBAT is an assessment tool that captures suicidal ideation, behavior, and risk. It permits assessment of change in suicidal ideation and behavior and documents clinician assessment of severity of suicidality and suicide risk. SIBAT is organized into 8 modules divided into 2 major divisions: patient-reported section (Modules 1-5) and clinician-rated section (Modules 6-8). Patient-reported section has modules of demographics and suicide history, risk/protective factors, suicidal thinking, suicide behavior, and suicide risk. Question 3 from Module 5 asks participants to describe their thinking about suicide right now from 5 response options ranging from 0 (I have no suicidal thoughts) to 4 (I have suicidal thoughts all of time). SIBAT Module 5 (My Risk) Question 3 (Patient-reported FoST) total score ranges from 0 to 4; a higher score indicates a more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline, Days 1, 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 1: number analyzed (Participants) | 111 | 110
  Change at Day 1 | 0.0 [-4 to 2] | 0.0 [-3 to 1]
  Change at Day 2: number analyzed (Participants) | 111 | 110
  Change at Day 2 | -1.0 [-4 to 1] | -1.0 [-4 to 2]
  Change at Day 4: number analyzed (Participants) | 110 | 108
  Change at Day 4 | -1.0 [-4 to 2] | -1.0 [-4 to 1]
  Change at Day 8: number analyzed (Participants) | 108 | 104
  Change at Day 8 | -1.0 [-4 to 1] | -1.0 [-4 to 1]
  Change at Day 11: number analyzed (Participants) | 103 | 100
  Change at Day 11 | -1.0 [-4 to 1] | -1.5 [-4 to 1]
  Change at Day 15: number analyzed (Participants) | 100 | 104
  Change at Day 15 | -1.0 [-4 to 1] | -2.0 [-4 to 1]
  Change at Day 18: number analyzed (Participants) | 94 | 101
  Change at Day 18 | -2.0 [-4 to 1] | -2.0 [-4 to 1]
  Change at Day 22: number analyzed (Participants) | 92 | 104
  Change at Day 22 | -2.0 [-4 to 2] | -2.0 [-4 to 1]
  Change at Day 25: number analyzed (Participants) | 93 | 96
  Change at Day 25 | -2.0 [-4 to 1] | -2.0 [-4 to 1]

15. Secondary Outcome: Change From Baseline in Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 7 - Clinician-rated FoST Total Score at Days 1, 2, 4, 8, 11, 15, 18, 22 and 25 During Double-blind Phase
Description: SIBAT is assessment tool that captures suicidal ideation, behavior, and risk. It permits assessment of change in suicidal ideation and behavior and documents clinician assessment of severity of suicidality and suicide risk. SIBAT has 8 modules divided into 2 major divisions: patient-reported section (Modules 1-5) and clinician-rated section (Modules 6-8). Clinician-rated section has modules for semi-structured interview, clinical global impressions of current severity of suicidality and imminent suicide risk, clinical global impression of long-term suicide risk, and clinical judgment of optimal suicide management. The score anchor point as in participant report frequency of suicidal thinking (FoST) that is, response options from never to all the time. Module 7-FoST score ranges from 0-5; higher score indicates more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline and Days 1, 2, 4, 8, 11, 15, 18, 22 and 25
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 112
units on a scale
  Change at Day 1: number analyzed (Participants) | 112 | 109
  Change at Day 1 | -1.0 [-5 to 2] | -1.0 [-5 to 1]
  Change at Day 2 | -1.0 [-5 to 1] | -1.0 [-5 to 1]
  Change at Day 4: number analyzed (Participants) | 110 | 109
  Change at Day 4 | -1.0 [-5 to 1] | -2.0 [-5 to 2]
  Change at Day 8: number analyzed (Participants) | 108 | 104
  Change at Day 8 | -2.0 [-5 to 2] | -2.0 [-5 to 1]
  Change at Day 11: number analyzed (Participants) | 102 | 100
  Change at Day 11 | -2.0 [-5 to 2] | -2.0 [-5 to 2]
  Change at Day 15: number analyzed (Participants) | 99 | 104
  Change at Day 15 | -2.0 [-5 to 0] | -2.0 [-5 to 1]
  Change at Day 18: number analyzed (Participants) | 94 | 102
  Change at Day 18 | -2.0 [-5 to 1] | -2.0 [-5 to 1]
  Change at Day 22: number analyzed (Participants) | 91 | 104
  Change at Day 22 | -2.0 [-5 to 1] | -2.0 [-5 to 1]
  Change at Day 25: number analyzed (Participants) | 93 | 95
  Change at Day 25 | -2.0 [-5 to 1] | -3.0 [-5 to 1]

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): DB Treatment Phase
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. A TEAE is categorized as related if assessed by the investigator as possibly, probably, or very likely related to study agent.
Time Frame: Up to Day 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants | 83 | 100

17. Secondary Outcome: Number of Participants With Treatment Emergent Abnormal Laboratory Values: DB Treatment Phase
Description: Low/high abnormal values are: Alanine aminotransferase (ALT)-high=200 Units per liter(U/L); ALP-high=250U/L; aspartate aminotransferase(AST)-high=250U/L; gamma glutamyl transferase(GGT)=300U/L; Albumin(low=24g/L,high=60 g/L); Bicarbonate(low=15.1, high=34.9mmol/L); Bilirubin(high=51.3micromol/L); calcium(low=1.5,high=3mmol/L);Chloride(low=94,high=112mmol/L); CK(High=990U/L); Creatinine(High=265.2micromol/L); Eosinophils(High=10%); Erythrocytes(low=3.0*1012/L,high=6.4*1012/L); Glucose(low=2.2,high=16.7mmol/L); Hemoglobin(low=80g/L,high=190g/L);Hematocrit(low=0.28, high=0.55 fraction); LD(high=500U/L); Leukocytes(low=2.5*109/L,high=15.5*109/L); Lymphocytes(low=10%,high=60%); Monocytes(high=20%); Neutrophils(low=30%,high=90%); Phosphate(low=0.7 mmol/L,high=2.6mmol/L); Platelet count(low=100*109/L,high=600*109/L]; Potassium(low=3.0mmol/L,high=5.8 mmol/L]; Protein(low=50 g/L); Sodium(low=125 mmol/L,high=155 mmol/L); Urate(low=89.2 micromol/L,high=594.8micromol/L); Urine(high=8.0 pH).
Time Frame: Up to Day 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase. Here 'n' (number analyzed) signifies number of participants analyzed for each specified category.ULN=upper limit of normal; mmol/L= millimoles per liter; micromol/L=micromole/liter; g/L=gram per liter
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants
  ALT>3*ULN: number analyzed (Participants) | 100 | 109
  ALT>3*ULN | 1 | 1
  ALT: Abnormal High: number analyzed (Participants) | 100 | 109
  ALT: Abnormal High | 1 | 1
  Albumin: Abnormal High: number analyzed (Participants) | 102 | 110
  Albumin: Abnormal High | 0 | 0
  Albumin: Abnormal Low: number analyzed (Participants) | 102 | 110
  Albumin: Abnormal Low | 0 | 0
  Alkaline phosphatase (ALP): Abnormal High: number analyzed (Participants) | 102 | 110
  Alkaline phosphatase (ALP): Abnormal High | 0 | 0
  AST: AST>3*ULN: number analyzed (Participants) | 100 | 108
  AST: AST>3*ULN | 0 | 0
  AST: Abnormal High: number analyzed (Participants) | 100 | 108
  AST: Abnormal High | 0 | 0
  Bicarbonate: Abnormal High: number analyzed (Participants) | 99 | 109
  Bicarbonate: Abnormal High | 0 | 0
  Bicarbonate: Abnormal Low: number analyzed (Participants) | 99 | 109
  Bicarbonate: Abnormal Low | 0 | 0
  Bilirubin: Abnormal High: number analyzed (Participants) | 100 | 109
  Bilirubin: Abnormal High | 0 | 0
  Calcium: Abnormal High: number analyzed (Participants) | 102 | 110
  Calcium: Abnormal High | 0 | 0
  Calcium: Abnormal Low: number analyzed (Participants) | 102 | 110
  Calcium: Abnormal Low | 0 | 0
  Chloride: Abnormal High: number analyzed (Participants) | 102 | 110
  Chloride: Abnormal High | 0 | 0
  Chloride: Abnormal Low: number analyzed (Participants) | 102 | 110
  Chloride: Abnormal Low | 0 | 0
  Creatine Kinase (CK): Abnormal High: number analyzed (Participants) | 100 | 109
  Creatine Kinase (CK): Abnormal High | 0 | 1
  Creatinine: Abnormal High: number analyzed (Participants) | 102 | 110
  Creatinine: Abnormal High | 0 | 0
  GGT: Abnormal High: number analyzed (Participants) | 102 | 110
  GGT: Abnormal High | 0 | 0
  Glucose: Abnormal High: number analyzed (Participants) | 100 | 109
  Glucose: Abnormal High | 0 | 0
  Glucose: Abnormal Low: number analyzed (Participants) | 100 | 109
  Glucose: Abnormal Low | 0 | 0
  ALT>3*ULN or AST>3*ULN and BILI>2*ULN: number analyzed (Participants) | 100 | 109
  ALT>3*ULN or AST>3*ULN and BILI>2*ULN | 0 | 0
  Lactate Dehydrogenase(LD): Abnormal High: number analyzed (Participants) | 94 | 101
  Lactate Dehydrogenase(LD): Abnormal High | 0 | 0
  Phosphate: Abnormal High: number analyzed (Participants) | 102 | 110
  Phosphate: Abnormal High | 0 | 0
  Phosphate: Abnormal Low: number analyzed (Participants) | 102 | 110
  Phosphate: Abnormal Low | 1 | 2
  Potassium: Abnormal High: number analyzed (Participants) | 102 | 110
  Potassium: Abnormal High | 0 | 0
  Potassium: Abnormal Low: number analyzed (Participants) | 102 | 110
  Potassium: Abnormal Low | 0 | 0
  Protein: Abnormal Low: number analyzed (Participants) | 102 | 110
  Protein: Abnormal Low | 0 | 0
  Sodium: Abnormal High: number analyzed (Participants) | 102 | 110
  Sodium: Abnormal High | 0 | 0
  Sodium: Abnormal Low: number analyzed (Participants) | 102 | 110
  Sodium: Abnormal Low | 0 | 0
  Urate: Abnormal High: number analyzed (Participants) | 102 | 110
  Urate: Abnormal High | 0 | 0
  Urate: Abnormal Low: number analyzed (Participants) | 102 | 110
  Urate: Abnormal Low | 0 | 0
  Basophils: Abnormal High: number analyzed (Participants) | 97 | 105
  Basophils: Abnormal High | 0 | 0
  Eosinophils: Abnormal High: number analyzed (Participants) | 97 | 105
  Eosinophils: Abnormal High | 0 | 0
  Erythrocytes: Abnormal High: number analyzed (Participants) | 97 | 105
  Erythrocytes: Abnormal High | 1 | 1
  Erythrocytes: Abnormal Low: number analyzed (Participants) | 97 | 105
  Erythrocytes: Abnormal Low | 0 | 0
  Hematocrit: Abnormal High: number analyzed (Participants) | 96 | 103
  Hematocrit: Abnormal High | 0 | 0
  Hematocrit: Abnormal Low: number analyzed (Participants) | 96 | 103
  Hematocrit: Abnormal Low | 0 | 0
  Hemoglobin(Hb): Abnormal High: number analyzed (Participants) | 97 | 105
  Hemoglobin(Hb): Abnormal High | 0 | 0
  Hemoglobin: Abnormal Low: number analyzed (Participants) | 97 | 105
  Hemoglobin: Abnormal Low | 0 | 0
  Leukocytes: Abnormal High: number analyzed (Participants) | 97 | 105
  Leukocytes: Abnormal High | 0 | 0
  Leukocytes: Abnormal Low: number analyzed (Participants) | 97 | 105
  Leukocytes: Abnormal Low | 1 | 0
  Lymphocytes: Abnormal High: number analyzed (Participants) | 97 | 105
  Lymphocytes: Abnormal High | 0 | 0
  Lymphocytes: Abnormal Low: number analyzed (Participants) | 97 | 105
  Lymphocytes: Abnormal Low | 0 | 0
  Monocytes: Abnormal High: number analyzed (Participants) | 97 | 105
  Monocytes: Abnormal High | 0 | 0
  Neutrophils: Abnormal High: number analyzed (Participants) | 97 | 105
  Neutrophils: Abnormal High | 0 | 0
  Neutrophils: Abnormal Low: number analyzed (Participants) | 97 | 105
  Neutrophils: Abnormal Low | 0 | 0
  Platelets: Abnormal High: number analyzed (Participants) | 97 | 104
  Platelets: Abnormal High | 0 | 0
  Platelets: Abnormal Low: number analyzed (Participants) | 97 | 104
  Platelets: Abnormal Low | 0 | 2
  Urine pH: Abnormal High: number analyzed (Participants) | 102 | 109
  Urine pH: Abnormal High | 0 | 0

18. Secondary Outcome: Number of Participants With Abnormal Nasal Examinations at Day 25: DB Treatment Phase
Description: Number of participants with abnormal nasal examination were reported. Nasal examination of visual inspection of the epistaxis, nasal crusts, nasal discharge, and nasal erythema was performed.
Time Frame: At Day 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase. Here, 'n' (number analyzed) signifies number of participants analyzed for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants
  Epistaxis: Mild: number analyzed (Participants) | 104 | 109
  Epistaxis: Mild | 0 | 1
  Epistaxis: Moderate: number analyzed (Participants) | 104 | 109
  Epistaxis: Moderate | 0 | 0
  Epistaxis: Severe: number analyzed (Participants) | 104 | 109
  Epistaxis: Severe | 0 | 0
  Nasal Crusts: Mild: number analyzed (Participants) | 104 | 109
  Nasal Crusts: Mild | 1 | 0
  Nasal Crusts: Moderate: number analyzed (Participants) | 104 | 109
  Nasal Crusts: Moderate | 0 | 0
  Nasal Crusts: Severe: number analyzed (Participants) | 104 | 109
  Nasal Crusts: Severe | 0 | 0
  Nasal Discharge: Mild: number analyzed (Participants) | 104 | 109
  Nasal Discharge: Mild | 0 | 3
  Nasal Discharge: Moderate: number analyzed (Participants) | 104 | 109
  Nasal Discharge: Moderate | 0 | 0
  Nasal Discharge: Severe: number analyzed (Participants) | 104 | 109
  Nasal Discharge: Severe | 0 | 0
  Nasal Erythema: Mild: number analyzed (Participants) | 104 | 109
  Nasal Erythema: Mild | 4 | 3
  Nasal Erythema: Moderate: number analyzed (Participants) | 104 | 109
  Nasal Erythema: Moderate | 0 | 0
  Nasal Erythema: Severe: number analyzed (Participants) | 104 | 109
  Nasal Erythema: Severe | 0 | 0

19. Secondary Outcome: Number of Participants With Treatment Emergent Abnormal Electrocardiogram (ECG) Values at Any Time: DB Treatment Phase
Description: Number of participants with treatment emergent abnormal ECG values for variables including heart rate (abnormally low refers to less than or equal to [<=] 50 beats per minute [bpm] , abnormally high refers greater than or equal to [>=] 100 bpm), pulse rate (PR) interval (abnormally high refers to >= 210 milliseconds [msec]), QRS interval (abnormally Low refers to <= 50, abnormally high refers to >= 120 msec) and QT interval (abnormally low refers to <= 200, abnormally high >= 500 msec) were reported.
Time Frame: Up to Day 25
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants
  Heart Rate <= 50 bpm | 8 | 2
  Heart Rate >= 100 bpm | 4 | 5
  PR Duration >= 210 msec | 3 | 5
  QRS Duration <= 50 msec | 0 | 0
  QRS Duration >= 120 msec | 0 | 0
  QT Duration <= 200 msec | 0 | 0
  QT Duration >= 500 msec | 0 | 0

20. Secondary Outcome: Number of Participants With Abnormal Arterial Oxygen Saturation (SpO2) Levels (Less Than [<] 93%) as Assessed by Pulse Oximetry at Any Time: DB Treatment Phase
Description: Pulse oximetry was used to measure arterial SpO2 levels. On each dosing day, the device was attached to the finger, toe, or ear, and SpO2 was monitored and documented. If oxygen saturation levels were less than (<) 93% at any time during the 1.5 hours postdose interval, pulse oximetry was recorded every 5 minutes until levels return to >= 93% or until the participant is referred for appropriate medical care, if clinically indicated. Participants with at least 2 consecutive postdose oxygen saturation below 93% during the DB treatment phase were reported.
Time Frame: Up to Day 25
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants | 2 | 1

21. Secondary Outcome: Number of Participants With Treatment Emergent Vital Signs Abnormalities: DB Treatment Phase
Description: Number of participants with treatment emergent vital signs abnormalities (pulse rate in bpm [abnormally low = a decrease from baseline of >= 15 to a value <= 50; abnormally high = an increase from baseline of >=15 to a value >=100] , systolic blood pressure [SBP] in mmHg [abnormally low = a decrease from baseline of >= 20 to a value <= 90; abnormally high = an increase from baseline of >= 20 to a value >= 180], and diastolic blood pressure [DBP] in mmHg [abnormally low= a decrease from baseline of >=15 to a value <= 50; abnormally high = an increase from baseline of >= 15 to a value >= 105) were reported.
Time Frame: Up to Day 25
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants
  Pulse rate (bpm): Decrease of >=15 to <=50 | 2 | 3
  Pulse rate (bpm): Increase of >=15 to >=100 | 6 | 13
  SBP (mmHg): Decrease of >=20 to <=90 | 4 | 0
  SBP (mmHg): Increase of >=20 to >=180 | 0 | 2
  DBP (mmHg): Decrease of >=15 to <=50 | 4 | 0
  DBP (mmHg): Increase of >=15 to >=105 | 1 | 11

22. Secondary Outcome: Number of Sedated Participants as Assessed by Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Score at Any Time: DB Treatment Phase
Description: MOAA/S was used to measure treatment-emergent sedation with correlation to levels of sedation defined by the American society of anesthesiologists (ASA) continuum. The MOAA/S scores range from 0 to 5 where,0 = no response to painful stimulus; ASA continuum = general anesthesia, 1 = responds to trapezius squeeze; ASA continuum = deep sedation, 2 = purposeful response to mild prodding or mild shaking; ASA continuum = moderate sedation, 3 = responds after name called loudly or repeatedly; ASA continuum = moderate sedation, 4 = lethargic response to name spoken in normal tone; ASA continuum = moderate sedation and 5 = readily responds to name spoken in normal tone (awake); ASA continuum = minimal sedation.
Time Frame: Up to Day 25
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants
  Score <=2: Yes | 0 | 3
  Score <=3: Yes | 1 | 13
  Score <=4: Yes | 20 | 43

23. Secondary Outcome: Number of Participants With an Increase in Clinician-administered Dissociative States Scale (CADSS) Total Score Over Time: DB Treatment Phase
Description: The CADSS used to measure present-state dissociative symptoms, and to assess treatment-emergent dissociative symptoms. It comprises 23 subjective items divided into 3 components: depersonalization (with score range from 0 to 28), derealization (with score range from 0 to 52), and amnesia (with score range from 0 to 8). Participants responses are coded on a 5-point scale (0 = "Not at all", 1 = "Mild", 2 = "Moderate", 3 = 'Severe" and 4 = "Extreme"). The total score is sum of the 23 items and range from 0 to 92, where 0 (best) and 92 (worst). A higher score indicates a more severe condition. Number of participants with an increase in CADSS total score (increase based on maximum CADSS total score change from predose of > 0) was reported.
Time Frame: Days 1, 4, 8, 11, 15, 18, 22 and 25
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug in the DB treatment phase. Here, 'n' (number analyzed) signifies the number of participants analyzed for each specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
Number analyzed (Participants) | 112 | 113
Participants
  Day 1: number analyzed (Participants) | 111 | 113
  Day 1 | 34 | 95
  Day 4: number analyzed (Participants) | 107 | 106
  Day 4 | 23 | 84
  Day 8: number analyzed (Participants) | 108 | 108
  Day 8 | 29 | 81
  Day 11: number analyzed (Participants) | 101 | 100
  Day 11 | 19 | 77
  Day 15: number analyzed (Participants) | 97 | 105
  Day 15 | 17 | 69
  Day 18: number analyzed (Participants) | 92 | 102
  Day 18 | 19 | 70
  Day 22: number analyzed (Participants) | 93 | 102
  Day 22 | 16 | 70
  Day 25: number analyzed (Participants) | 91 | 98
  Day 25 | 14 | 72

ADVERSE EVENTS:
Time Frame: Up to Day 25
Description: Safety analysis set included all randomized participants who received at least 1 dose of study agent in the double-blind treatment phase.
Groups:
- Placebo Plus SOC Antidepressant Treatment: Subjects self-administered placebo matched to esketamine intranasally (1 spray of placebo to each nostril at 0, 5 and 10 minutes) twice per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25) plus received standard of care (SOC) antidepressant treatment which was initiated or optimized on Day 1 during double blind phase (DB).
- Esketamine 84 mg Plus SOC Antidepressant Treatment: Subjects self-administered esketamine 84 milligram (mg) intranasally (1 spray of esketamine 14 mg to each nostril at 0, 5 and 10 minutes) twice per week for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25) plus received SOC antidepressant treatment which was initiated or optimized on Day 1 during double blind phase.
Arm/Group | Placebo Plus SOC Antidepressant Treatment | Esketamine 84 mg Plus SOC Antidepressant Treatment
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/113
Serious Adverse Events (participants affected / at risk) | 6/112 | 4/113
Other Adverse Events (participants affected / at risk) | 66/112 | 91/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus SOC Antidepressant Treatment (N=112) | Esketamine 84 mg Plus SOC Antidepressant Treatment (N=113)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Depression Suicidal (Psychiatric disorders) | 1 | 2
Suicidal Ideation (Psychiatric disorders) | 2 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus SOC Antidepressant Treatment (N=112) | Esketamine 84 mg Plus SOC Antidepressant Treatment (N=113)
Vertigo (Ear and labyrinth disorders) | 1 | 7
Vision Blurred (Eye disorders) | 5 | 10
Constipation (Gastrointestinal disorders) | 5 | 15
Nausea (Gastrointestinal disorders) | 15 | 23
Vomiting (Gastrointestinal disorders) | 7 | 8
Blood Pressure Increased (Investigations) | 6 | 19
Dizziness (Nervous system disorders) | 10 | 40
Dizziness Postural (Nervous system disorders) | 2 | 6
Dysgeusia (Nervous system disorders) | 11 | 16
Headache (Nervous system disorders) | 20 | 21
Hypoaesthesia (Nervous system disorders) | 2 | 8
Sedation (Nervous system disorders) | 2 | 7
Somnolence (Nervous system disorders) | 11 | 21
Anxiety (Psychiatric disorders) | 10 | 6
Dissociation (Psychiatric disorders) | 4 | 33
Insomnia (Psychiatric disorders) | 7 | 7

LIMITATIONS AND CAVEATS:
Esketamine's known characteristic effects such as dissociative symptoms, sedation, and elevation of blood pressure may have impact on blinding, to minimize this bias, protocol specified that different raters perform efficacy and safety assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03039192/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03039192/SAP_001.pdf